CLINICAL TRIAL: NCT05285839
Title: Single Center, Pilot Study to Evaluate the Effectiveness and Safety of Dupilumab in Combination With Narrowband UVB (nUVB) Phototherapy in the Treatment of Moderate-to-Severe Atopic Dermatitis
Brief Title: Dupixent and Narrowband UVB for Atopic Dermatitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Psoriasis Treatment Center of Central New Jersey (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETC01
Record Dates: First submitted 2022-03-08; First posted 2022-03-18 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dupixent and Narrowband UVB (Experimental): Dupixent and Narrowband UVB
  Interventions: Drug: Dupixent

INTERVENTIONS:
Drug: Dupixent — dupilumab 300mg

SUMMARY:
24 weeks open-label study with dupilumab and narrowband UVB phototherapy three times weekly for 12 weeks followed by 12 weeks of dupilumab monotherapy.

DETAILED DESCRIPTION:
24 weeks open-label study with dupilumab and narrowband UVB phototherapy three times weekly for 12 weeks followed by 12 weeks of dupilumab monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adult ≥ 18 years of age;
* Diagnosis of moderate to severe atopic dermatitis as defined at baseline by:

  * EASI score of 16 or greater,
  * IGA score of 3 or greater
  * BSA of 10% or greater,

Exclusion Criteria:

* Subjects with previous exposure to dupilumab.
* Known or suspected hypersensitivity to dupilumab or any of its excipients.
* History of photosensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Investigators Global Assessment Score of score of 0 or 1 | 12 weeks
  Proportion of subjects achieving an IGA score of 0 or 1 with at least a 2 grade improvement at week 12

CONTACTS AND LOCATIONS:
Locations (1):
- Eczema Treatment Center of New Jersey, East Windsor, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No